CLINICAL TRIAL: NCT00765102
Title: A Phase II Trial of Romidepsin and Bortezomib for Multiple Myeloma Patients With Relapsed or Refractory Disease
Brief Title: Trial of Romidepsin and Bortezomib for Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: There was a change in the Sponsor's research strategy; safety concerns were not a factor.
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GPI-08-0006
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Results first posted 2012-12-20 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myelonoma; Romidepsin; Bortezomib
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; romidepsin; Depsipeptides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Romidepsin + Bortezomib (Experimental): Romidepsin was given as an infusion on Days 1, 8 and 15 of each 28-day cycle. Bortezomib was administered twice a week for two consecutive weeks (Days 1, 4, 8 and 11) followed by a 17-day rest period.
  Patients were treated to a maximum response plus two additional cycles or a maximum of eight cycles.
  Interventions: Drug: Bortezomib; Drug: Romidepsin

INTERVENTIONS:
Drug: Bortezomib — Bortezomib was administered at a dose of 1.0 mg/m^2 as an intravenous (IV) push over 3 to 5 seconds twice weekly for 2 consecutive weeks (Days 1, 4, 8 and 11) of each 28-day cycle. On days that bortezomib and romidepsin were administered together, bortezomib was administered prior to the romidepsin infusion.
  Patients were treated to a maximum response plus two additional cycles or a maximum of eight cycles.
  Other Names: VELCADE®
Drug: Romidepsin — Romidepsin initially was administered at a dose of 10 mg/m^2 as a 1-hour intravenous (IV) infusion on Days 1, 8, and 15 of each 28-day cycle. Based on the occurrence of Grade 3 thrombocytopenia at this dose level, the dose was reduced by protocol amendment to 8 mg/m^2.
  Other Names: ISTODAX®; depsipeptide; FK228

SUMMARY:
This is a phase II, open-label, multicenter, dual-strata study designed to evaluate the efficacy and safety of IV romidepsin given in combination with IV bortezomib for multiple myeloma (MM) patients with refractory or relapsed disease. Patients will be enrolled into one of two strata, bortezomib-resistant or bortezomib non-resistant.

ELIGIBILITY:
Inclusion Criteria

Patients must fulfill all of the following criteria to be eligible for study participation:

* Male or female patients aged ≥ 18 years old
* Has given voluntary written informed consent before any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care
* Previously diagnosed with multiple myeloma (MM) based on standard criteria as follows:

  * Major criteria:

    1. Plasmacytomas on tissue biopsy.
    2. Bone marrow plasmacytosis (>30% plasma cells).
    3. Monoclonal immunoglobulin spike on serum electrophoresis IgG >3.5 g/dL or IgA >2.0 g/dL; kappa or lambda light chain excretion >1 g/day on 24 hour urine protein electrophoresis
  * Minor criteria:

    1. Bone marrow plasmacytosis (10 to 30% plasma cells)
    2. Monoclonal immunoglobulin present but of lesser magnitude than given under major criteria
    3. Lytic bone lesions.
    4. Normal IgM <50 mg/dL, IgA <100 mg/dL or IgG <600 mg/dL

Any of the following sets of criteria will confirm the diagnosis of MM:

* Any two of the major criteria
* Major criterion 1 plus minor criterion 2, 3, or 4.
* Major criterion 3 plus minor criterion 1 or 3.
* Minor criteria 1, 2, and 3 or 1, 2, and 4.
* Currently has MM with:

  o Measurable disease, defined as a monoclonal immunoglobulin spike on serum electrophoresis of >=1 gm/dL and/or urine monoclonal immunoglobulin spike of >=200 mg/24 hours, or evidence of lytic bone disease
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* Life-expectancy > 3 months
* All women of childbearing potential must use an effective barrier method of contraception. Male patients should use a barrier method of contraception during the treatment period and for 3 months thereafter
* Patients must meet the following laboratory criteria at Baseline (Day 1 of Cycle 1, before study drug administration):

  * Platelet count ≥ 100*10^9/L
  * Absolute neutrophil count ≥ 1.5*10^9/L
  * OR if the bone marrow is extensively infiltrated
  * Platelet count ≥ 75*10^9/L
  * Absolute neutrophil count ≥ 1.0*10^9/L
* Patients must meet the following laboratory criteria at the Screening visit conducted within 14 days of enrollment (Day 1, Cycle 1):

  * o Aspartate transaminase/serum glutamic oxaloacetic transaminase (AST/SGOT) and alanine transaminase/serum glutamic pyruvic transaminase (ALT/SGPT) ≤ 3.0*upper limit of normal (ULN)
  * Serum bilirubin ≤ 2.0*ULN
  * Calculated or measured creatinine clearance: ≥30 mL/minute. Patient with a creatinine >10mL/min and <30 mL/min due to significant myelomatous involvement of the kidneys may be enrolled in the study after receipt of approval from the lead investigator and sponsor
  * Serum potassium ≥ 3.8 mmol/L
  * Serum magnesium >1.8 mg/dL
  * Serum phosphorus ≥ lower limit of normal (LLN)

Exclusion Criteria

Patients are ineligible for entry if any of the following criteria are met:

* Chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) or thalidomide, lenalidomide, arsenic trioxide, bortezomib, or glucocorticosteroids within 3 weeks prior to the first dose of romidepsin
* Prior major surgery within 3 weeks prior to the first day of treatment
* Use of any investigational agent within 4 weeks of study entry
* Prior therapy with romidepsin
* Any known cardiac abnormalities such as:

  * Congenital long QT syndrome;
  * QTc interval ≥ 500 milliseconds;
  * Myocardial infarction within 6 months of Day 1. Subjects with a history of myocardial infarction between 6 and 12 months prior to the first day of cycle one who are asymptomatic and have had a negative cardiac risk assessment (treadmill stress test, nuclear medicine stress test, or stress echocardiogram) since the event may participate;
  * Other significant electrocardiogram (ECG) abnormalities including 2nd degree atrio-ventricular (AV) block type II, 3rd degree AV block, or bradycardia (ventricular rate less than 50 beats/min);
  * Symptomatic coronary artery disease (CAD), e.g., angina Canadian Class II-IV In any patient in whom there is doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present;
  * An ECG recorded at screening showing evidence of cardiac ischemia (ST depression depression of ≥2 mm, measured from isoelectric line to the ST segment). If in any doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present;
  * Congestive heart failure (CHF) that meets New York Heart Association (NYHA) Class II to IV definitions and/or ejection fraction <40% by Multi Gated Acquisition Scan (MUGA scan) or <50% by echocardiogram and/or MRI;
  * A known history of sustained ventricular tachycardia (VT), ventricular fibrillation (VF), Torsade de Pointes, or cardiac arrest unless currently addressed with an automatic implantable cardioverter defibrillator (AICD);
  * Hypertrophic cardiomegaly or restrictive cardiomyopathy from prior treatment or other causes;
  * Uncontrolled hypertension, i.e., blood pressure (BP) of ≥160/95; patients who have a history of hypertension controlled by medication must be on a stable dose (for at least one month) and meet all other inclusion criteria; or
  * Any cardiac arrhythmia requiring an anti-arrhythmic medication (excluding stable doses of beta-blockers)
* POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein (M-protein) and skin changes)
* Plasma cell leukemia
* Primary amyloidosis
* Patients with a prior malignancy within the last 5 years (except for basal or squamous cell carcinoma, or in situ cancer of the cervix)
* Severe hypercalcemia, i.e., serum calcium ≥14 mg/dL (3.5 mmol/L)
* Known infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* Other concurrent severe and/or uncontrolled medical or psychiatric conditions.
* Concomitant use of drugs that may cause a prolongation of the QTc
* Concomitant use of CYP3A4 inhibitors
* Patients who have hypersensitivity to bortezomib, boron or mannitol
* Patients who are pregnant or breast-feeding
* Patients with any significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to him/her by the study staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-09-01 (Actual); Primary Completion 2010-03-01 (Actual); Study Completion 2010-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tina Neilson, Study Director — Celgene Corporation
Locations (12):
- United States (12):
  - Loma Linda University Cancer Center, Loma Linda, California
  - Desert Cancer Care, Inc, Rancho Mirage, California
  - Santa Barbara Hematology Oncology Medical Group, Inc., Santa Barbara, California
  - James R Berenson, MD, Inc., West Hollywood, California
  - Georgia Cancer Specialists I, PC, Atlanta, Georgia
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Mecklenburg Medical Group, Charlotte, North Carolina
  - Baylor Sammons Cancer Center, Dallas, Texas
  - Dallas Oncology Consultants, P.A., Duncanville, Texas
  - Oncology Consultants, P.A, Houston, Texas
  - Central Utah Clinic, PC, Provo, Utah
  - Virginia Mason Medical Centre, Seattle, Washington

REFERENCES:
- [Background] Berenson J, et al. A phase II study of a 1-hour infusion of romidepsin combined with bortezomib for multiple myeloma (MM) patients with relapsed or refractory disease. Presented at 2009 ASCO Annual Meeting, May 29-June 2, 2009, Orlando FL. Abstract No. e10908. J Clin Oncol 2009;27(15s)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Stratum 1 (bortezomib resistant) had 19 participants. Stratum 2 (non-bortezomib resistant) had 13 participants.
Period: Overall Study
Arm/Group | Romidepsin + Bortezomib
Started | 32
Completed | 1 (Completed 8 cycles of treatment)
Not Completed | 31
Not completed — Progressive disease | 18
Not completed — Adverse Event | 6
Not completed — Physician Decision | 4
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Romidepsin + Bortezomib
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (8.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 14
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 2
  White | 24
  Other | 2
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is a scale that measures how cancer affects a patient. The scale ranges from 0 (fully active) to 5 (dead). 0=Fully active without restriction; 1= Restricted in physically strenuous activity; 2= Ambulatory, capable of all selfcare.
  participants
    Status 0 | 12
    Status 1 | 14
    Status 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Count of Participant Best Overall Response As Assessed by the Investigator
Description: Complete Response: disappearance of monoclonal protein from blood and urine, and disappearance of soft tissue plasmacytomas, <5% plasmas cells in marrow and no increase of lytic bone lesions.
  Very Good Partial Response: disappearance of plasmacytomas, no increase of lytic bone lesions, serum and urine M-protein not detectable by immunofixation, other.
  Partial Response: >=50% decrease in serum monoclonal protein, and in soft tissue plasmacytomas, no increase of lytic bone lesions, other.
  Minimal Response (MR): ≥ 25% to ≤ 49% decrease in serum monoclonal protein, and in size of plasmacytomas, no increase of lytic bone lesions, other.
  Stable Disease: Less than MR, but not PD
  Progressive Disease(PD):>25% increase in serum monoclonal paraprotein, or >25% plasma cells in marrow, or >25% increase in 24-hour urinary light chain excretion or increase in existing lytic bone lesions or soft tissue plasmacytomas or new bone lesions or soft tissue plasmacytomas, or hypercalcemia.
Time Frame: up to 8 months
Population: Intent-to-Treat (ITT) population of patients defined as all patients who receive at least one dose of romidepsin and bortezomib. However efficacy data was not analyzed due to the early termination of the study.
Arm/Group | Romidepsin + Bortezomib
Number analyzed (Participants) | 0

2. Secondary Outcome: Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Counts of participants with TEAEs, and subset by relation to drug, grade of severity, serious, TEAEs leading to discontinuation or leading to death. AEs were graded for severity according to the National Cancer Institute Common Terminology Criteria (NCI CTCAE), V 3.0: Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe (prevents normal everyday activities); Grade 4: Life-threatening or disabling; Grade 5: Death.
Time Frame: up to 9 months
Population: Safety population of participants who took at least one dose of drug.
Measure: Number; unit: participants
Arm/Group | Romidepsin + Bortezomib
Number analyzed (Participants) | 32
participants
  At least 1 TEAE | 32
  At least 1 drug-related TEAE | 30
  At least 1 Romidepsin-related TEAE | 28
  At least 1 Bortezomib-related TEAE | 30
  At least 1 >=Grade 3 TEAE | 28
  At least 1 Grade 4 TEAE | 5
  At least 1 serious TEAE | 14
  At least 1 TEAE leading to discontinuation | 6
  At least 1 TEAE leading to death | 2

3. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-∞)
Description: AUC (0 - ∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞) of Romidepsin based on plasma samples.
Time Frame: Day 1 (cycle 1): 1 hour prior to romidepsin administration, 0.25, 0.5, 1, 2, 3, 4, 6, and 24 hours after initiation of romidepsin infusion
Population: A subset of participants from the lead investigator's site had PK samples taken.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Romidepsin 8 mg/m^2 + Bortezomib: Each patient enrolled in the PK portion underwent one PK sampling period on Day 1 of Cycle 1, following the administration of Bortezomib and 1-hour IV infusion of romidepsin 8mg/m^2.
- Romidepsin 10 mg/m^2 + Bortezomib: Each patient enrolled in the PK portion underwent one PK sampling period on Day 1 of Cycle 1, following the administration of Bortezomib and 1-hour IV infusion of romidepsin 10mg/m^2.
Arm/Group | Romidepsin 8 mg/m^2 + Bortezomib | Romidepsin 10 mg/m^2 + Bortezomib
Number analyzed (Participants) | 6 | 5
ng*hr/mL | 1209.1 (29.4) | 1149.5 (22.2)

4. Secondary Outcome: Maximum Observed Concentration (Cmax)
Description: Maximum observed concentration of Romidepsin
Time Frame: as for outcome 3
Population: A subset of participants from the lead investigator's site had PK samples taken.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Romidepsin 8 mg/m^2 + Bortezomib | Romidepsin 10 mg/m^2 + Bortezomib
Number analyzed (Participants) | 6 | 5
ng/mL | 913.9 (21.4) | 1002.7 (20.6)

5. Secondary Outcome: Time to Maximum Observed Concentration (Tmax)
Description: Time to maximum observed concentration of Romidepsin
Time Frame: as for outcome 3
Population: A subset of participants from the lead investigator's site had PK samples taken.
Measure: Median (Full Range); unit: hr
Arm/Group | Romidepsin 8 mg/m^2 + Bortezomib | Romidepsin 10 mg/m^2 + Bortezomib
Number analyzed (Participants) | 6 | 5
hr | 1.04 [0.60 to 1.10] | 0.58 [0.53 to 0.67]

6. Secondary Outcome: Terminal Half-life (t1/2)
Description: Terminal half-life of Romidepsin
Time Frame: as for outcome 3
Population: A subset of participants from the lead investigator's site had PK samples taken.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Romidepsin 8 mg/m^2 + Bortezomib | Romidepsin 10 mg/m^2 + Bortezomib
Number analyzed (Participants) | 6 | 5
hr | 4.1 (11.0) | 3.6 (41.7)

7. Secondary Outcome: Total Clearance (CL)
Description: Total clearance of Romidepsin
Time Frame: as for outcome 3
Population: A subset of participants from the lead investigator's site had PK samples taken.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Romidepsin 8 mg/m^2 + Bortezomib | Romidepsin 10 mg/m^2 + Bortezomib
Number analyzed (Participants) | 6 | 5
L/hr | 11.3 (26.9) | 16.4 (31.5)

8. Secondary Outcome: Total Volume of Distribution (Vz)
Description: Total volume of distribution of Romidepsin
Time Frame: as for outcome 3
Population: A subset of participants from the lead investigator's site had PK samples taken.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Romidepsin 8 mg/m^2 + Bortezomib | Romidepsin 10 mg/m^2 + Bortezomib
Number analyzed (Participants) | 6 | 5
L | 66.5 (23.4) | 85.9 (66.8)

9. Secondary Outcome: Kaplan Meier Estimate for Time to Progression Assessed by the Investigator
Description: Time to progression of disease is defined as the time from initiation of therapy to progressive disease as assessed by the investigator.
  Progressive Disease(PD):>25% increase in serum monoclonal paraprotein, or >25% plasma cells in marrow, or >25% increase in 24-hour urinary light chain excretion or increase in existing lytic bone lesions or soft tissue plasmacytomas or new bone lesions or soft tissue plasmacytomas, or hypercalcemia.
  Disease progression for participants relapsing from a complete response: reappearance of serum or urinary paraprotein on imunofixation, >= 5% plasma cells in the bone marrow aspirate or biopsy, increase in existing lytic bone lesions or soft tissue plasmacytomas or new bone lesions or soft tissue plasmacytomas, development of hypercalcemia.
Time Frame: up to month 8
Population: Intent to treat population. Analysis was not performed due to early termination of the study.
Arm/Group | Romidepsin + Bortezomib
Number analyzed (Participants) | 0

10. Secondary Outcome: Kaplan Meier Estimate for Time to Response Assessed by the Investigator
Description: The time to the first response is defined as the time from the initiation of therapy to the first evidence of a confirmed response (complete response, very good partial response, partial response or minimal response).
  Complete Response: disappearance of monoclonal protein from blood and urine, and disappearance of soft tissue plasmacytomas, <5% plasmas cells in marrow and no increase of lytic bone lesions.
  Very Good Partial Response: disappearance of plasmacytomas, no increase of lytic bone lesions, serum and urine M-protein not detectable by immunofixation, other.
  Partial Response: >=50% decrease in serum monoclonal protein, and in soft tissue plasmacytomas, no increase of lytic bone lesions, other.
  Minimal Response (MR): ≥ 25% to ≤ 49% decrease in serum monoclonal protein, and in size of plasmacytomas, no increase of lytic bone lesions, other.
Time Frame: up to month 8
Population: Intent to treat population. However efficacy data was not analyzed due to the early termination of the study.
Arm/Group | Romidepsin + Bortezomib
Number analyzed (Participants) | 0

11. Secondary Outcome: Kaplan Meier Estimate for Duration of Response Assessed by the Investigator
Description: Duration of response is defined as the time from first response to progressive disease as assessed by the investigator.
  Progressive Disease(PD):>25% increase in serum monoclonal paraprotein, or >25% plasma cells in marrow, or >25% increase in 24-hour urinary light chain excretion or increase in existing lytic bone lesions or soft tissue plasmacytomas or new bone lesions or soft tissue plasmacytomas, or hypercalcemia.
  Disease progression for participants relapsing from a complete response: reappearance of serum or urinary paraprotein on imunofixation, >= 5% plasma cells in the bone marrow aspirate or biopsy, increase in existing lytic bone lesions or soft tissue plasmacytomas or new bone lesions or soft tissue plasmacytomas, development of hypercalcemia.
Time Frame: up to month 8
Population: Intent to treat population. However efficacy data was not analyzed due to the early termination of the study.
Arm/Group | Romidepsin + Bortezomib
Number analyzed (Participants) | 0

12. Secondary Outcome: Kaplan Meier Estimates for Progression-free Survival Assessed by the Investigator
Description: Progression-free survival is the time from initiation of therapy to progressive disease, removal from study for any reason, death from any cause, or the last follow-up visit, whichever occurs first.
  Progressive Disease(PD):>25% increase in serum monoclonal paraprotein, or >25% plasma cells in marrow, or >25% increase in 24-hour urinary light chain excretion or increase in existing lytic bone lesions or soft tissue plasmacytomas or new bone lesions or soft tissue plasmacytomas, or hypercalcemia.
  Disease progression for participants relapsing from a complete response: reappearance of serum or urinary paraprotein on imunofixation, >= 5% plasma cells in the bone marrow aspirate or biopsy, increase in existing lytic bone lesions or soft tissue plasmacytomas or new bone lesions or soft tissue plasmacytomas, development of hypercalcemia.
Time Frame: up to month 8
Population: Intent to treat population. However efficacy data was not analyzed due to the early termination of the study.
Arm/Group | Romidepsin + Bortezomib
Number analyzed (Participants) | 0

13. Secondary Outcome: Kaplan Meier Estimates for Overall Survival
Description: Overall survival is the time from initiation of therapy to death from any cause.
Time Frame: up to month 8
Population: Intent to treat population. However efficacy data was not analyzed due to the early termination of the study.
Arm/Group | Romidepsin + Bortezomib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: up to 9 months
Arm/Group | Romidepsin + Bortezomib
Serious Adverse Events (participants affected / at risk) | 14/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Romidepsin + Bortezomib (N=32)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 2
Pyrexia (General disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Pneumonia (Infections and infestations) | 2
Pneumonia primary atypical (Infections and infestations) | 1
Pneumonia staphylococcal (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Septic shock (Infections and infestations) | 2
Urosepsis (Infections and infestations) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 2
Electrocardiogram T wave inversion (Investigations) | 1
Electrocardiogram QT prolongation (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Renal failure acute (Renal and urinary disorders) | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
Venous thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Romidepsin + Bortezomib (N=32)
Anaemia (Blood and lymphatic system disorders) | 13
Leukopenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 21
Abdominal pain (Gastrointestinal disorders) | 2
Aphthous stomatitis (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 10
Diarrhoea (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 9
Asthenia (General disorders) | 2
Fatigue (General disorders) | 14
Infusion site erythema (General disorders) | 2
Malaise (General disorders) | 2
Oedema peripheral (General disorders) | 3
Pain (General disorders) | 2
Pyrexia (General disorders) | 8
Sinusitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 4
White blood cell count decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 4
Hyponatraemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 10
Neuropathy (Nervous system disorders) | 3
Neuropathy peripheral (Nervous system disorders) | 2
Renal failure (Renal and urinary disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash macular (Skin and subcutaneous tissue disorders) | 2
Flushing (Vascular disorders) | 2
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Upon investigator submission of a publication or presentation to Celgene, Celgene shall complete its review within 60 days after receipt of the proposed publication or presentation. Upon Celgene's request, proposed publication or presentation will be delayed up to 60 additional days to enable Celgene to secure adequate intellectual property protection of property of Celgene that would be affected by such proposed publication or presentation